CLINICAL TRIAL: NCT06938360
Title: Clinical Efficacy and Safety Assessment of Breast-Conserving Surgery for Central Breast Cancer: A Prospective Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Shaanxi Provincial People's Hospital (Other); Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20242433-F-1
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: breast-conserving surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: This study enrolled 158 patients with primary central early-stage breast cancer and randomly assigned them to two groups. The control group underwent total mastectomy (with optional prosthetic implantation or autologous tissue reconstruction), while the experimental group received breast-conserving surgery combined with radiotherapy (nipple resection with concurrent nipple reconstruction and oncoplastic surgery when nipple involvement was present; conversion to total mastectomy required for intraoperative or postoperative positive margins).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total mastectomy (with optional prosthetic implantation or autologous tissue reconstruction) (No Intervention): Prosthetic implantation or autologous tissue transfer reconstruction was permitted
- breast-conserving surgery combined with radiotherapy (Experimental): nipple resection with concurrent nipple reconstruction and oncoplastic surgery when nipple involvement was present; conversion to total mastectomy required for intraoperative or postoperative positive margins
  Interventions: Procedure: breast-conserving surgery combined with radiotherapy

INTERVENTIONS:
Procedure: breast-conserving surgery combined with radiotherapy — The experimental group received breast-conserving surgery combined with radiotherapy
  Arms: breast-conserving surgery combined with radiotherapy

SUMMARY:
This study enrolled 158 patients with primary central early-stage breast cancer and randomly assigned them to two groups. The control group underwent total mastectomy (with optional prosthetic implantation or autologous tissue reconstruction), while the experimental group received breast-conserving surgery combined with radiotherapy (nipple resection with concurrent nipple reconstruction and oncoplastic surgery when nipple involvement was present; conversion to total mastectomy required for intraoperative or postoperative positive margins). The primary endpoint was local recurrence rate, with secondary endpoints including disease-free survival (DFS), overall survival (OS), patient-reported outcomes (PRO), and surgery-related complications.

DETAILED DESCRIPTION:
This prospective, open-label, multicenter, randomized clinical trial plans to enroll 158 patients with primary central early-stage breast cancer. Participants will be randomly assigned to two groups: the control group undergoing total mastectomy (with optional prosthetic implantation or autologous tissue reconstruction), and the experimental group receiving breast-conserving surgery with radiotherapy (nipple resection with concurrent nipple reconstruction and oncoplastic surgery when nipple involvement is present; conversion to total mastectomy required for intraoperative or postoperative positive margins). All enrolled patients will initiate surgical treatment within 24 hours after eligibility confirmation. Experimental group patients must complete preoperative breast ultrasound, mammography, and MRI to assess breast-conserving feasibility. All patients receive standardized adjuvant therapy (chemotherapy, endocrine therapy, targeted therapy, and immunotherapy) according to guidelines. Those meeting neoadjuvant therapy criteria may receive preoperative systemic treatments (chemotherapy, endocrine therapy, targeted therapy, and immunotherapy), excluding neoadjuvant radiotherapy.

Primary Endpoint:

local recurrence rate

Secondary Endpoints:

disease-free survival (DFS), overall survival (OS), patient-reported outcomes (PRO), and surgery-related complications.

Inclusion Criteria:

1. Female patients aged 18-70 years with primary breast cancer;
2. Histopathologically confirmed invasive breast cancer (meeting latest ASCO/CAP guidelines criteria) with:

   * TNM stage T1-2;
   * Nodal stage N0-1;
3. Ductal carcinoma in situ (DCIS) with maximum tumor diameter <3 cm;
4. Paget's disease;
5. Neoadjuvant chemotherapy permitted for eligible patients;
6. Unicentric lesion confirmed by breast ultrasound, mammography, and MRI;
7. Nipple-areolar complex resection required for preoperative imaging or pathologically confirmed nipple involvement;
8. Enrolled patients randomized 1:1 to breast-conserving surgery or total mastectomy group;
9. Participants voluntarily signed informed consent forms and completed ethics review procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-70 years with primary breast cancer;
2. Histopathologically confirmed invasive breast cancer (meeting latest ASCO/CAP guidelines criteria) with:

   * TNM stage T1-2;
   * Nodal stage N0-1;
3. Ductal carcinoma in situ (DCIS) with maximum tumor diameter <3 cm;
4. Paget's disease;
5. Neoadjuvant chemotherapy permitted for eligible patients;
6. Unicentric lesion confirmed by breast ultrasound, mammography, and MRI;
7. Nipple-areolar complex resection required for preoperative imaging or pathologically confirmed nipple involvement;
8. Enrolled patients randomized 1:1 to breast-conserving surgery or total mastectomy group;
9. Participants voluntarily signed informed consent forms and completed ethics review procedures.

Exclusion Criteria:

1. Tumor-related characteristics

   1. Metastatic or bilateral breast cancer
   2. Inflammatory breast cancer
   3. Multicentric lesions
2. Comorbidities/treatment history

   1. History of other malignancies (except cured cervical carcinoma in situ/basal cell carcinoma/squamous cell carcinoma) or prior anticancer therapy (systemic/local)
   2. Major non-breast surgery within 4 weeks before enrollment (excluding diagnostic biopsy/PICC placement) without full recovery
   3. Active infections/immune disorders:

      HIV/AIDS Viral hepatitis (HBV-DNA≥500 IU/ml; HCV antibody-positive with detectable HCV-RNA) Autoimmune hepatitis HBV/HCV coinfection
   4. Allogeneic bone marrow/solid organ transplantation history or planned
   5. Cardiovascular diseases:

      * Heart failure or LVEF<50%
      * Uncontrolled arrhythmias (resting heart rate>100 bpm, ventricular tachycardia, Mobitz II/third-degree AV block)
      * Angina requiring antianginal drugs
      * Clinically significant valvulopathy
      * Transmural myocardial infarction on ECG
      * Uncontrolled hypertension (SBP>180 mmHg and/or DBP>100 mmHg)
3. Reproductive status

   Pregnancy/lactation, or reproductive-aged women with:
   * Positive baseline pregnancy test
   * Refusal of effective contraception
4. Neuropsychiatric disorders Epilepsy, dementia, psychoactive substance abuse, or alcoholism
5. Other investigator-determined exclusionary conditions

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2028-02-20 (Estimated); Study Completion 2030-02-20 (Estimated)

PRIMARY OUTCOMES:
Local recurrence rate (LRR) | From enrollment to 3 years later or death
  Local recurrence rate (LRR) was defined as tumor recurrence in the ipsilateral breast, chest wall, skin, or surgical scar area.

SECONDARY OUTCOMES:
Disease-free survival (DFS) | From enrollment to 3 years later or death
  Disease-free survival (DFS) was defined as the time from randomization to the first occurrence of any of the following events: ipsilateral/contralateral breast cancer recurrence; local/regional recurrence; distant metastasis; or all-cause death.
Overall survival (OS) | From enrollment to 3 years later or death
  Overall survival (OS) was defined as the time interval from enrollment to all-cause death.
Patient-reported outcomes (PRO) | From enrollment to 3 years later
  Patient-reported outcomes (PRO) were assessed using the BREAST-Q Cosmetic Module, with scores ranging from 0 to 100 (higher scores indicating better cosmetic outcomes).

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided